CLINICAL TRIAL: NCT00929188
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-42160443 as Adjunctive Therapy in Subjects With Cancer-Related Pain, Followed by an Open-Label Extension Phase
Brief Title: A Study of the Safety and Effectiveness of JNJ-42160443 as add-on Treatment in Patients With Cancer-related Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016057; 42160443PAI2001 (Other: Janssen Research & Development, LLC); 2008-007690-21 (EudraCT Number)
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Pain, Burning; Pain, Crushing; Pain, Migratory; Pain, Radiating; Pain, Splitting
Keywords: Moderate to severe chronic, cancer-related pain related to an active cancer; Cancer-related pain; Moderate to severe chronic pain; JNJ-42160443
MeSH Terms: conditions — Pain; Cancer Pain | interventions — fulranumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 (Experimental): JNJ-42160443 Type=1 unit=mg number=10 form=solution for injection route=subcutaneous use. SC injection (10mg/ml) once every 4 weeks for up to 52 weeks
  Interventions: Drug: JNJ-42160443
- 002 (Placebo Comparator): Placebo Form=solution for injection route=subcutaneous use. SC injection (0.9 mL matching placebo) once on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42160443 — Type=1, unit=mg, number=10, form=solution for injection , route=subcutaneous use. SC injection (10mg/ml) once every 4 weeks for up to 52 weeks
  Arms: 001
Drug: Placebo — Form=solution for injection, route=subcutaneous use. SC injection (0.9 mL matching placebo) once on Day 1
  Arms: 002

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of JNJ-42160443 with placebo in the treatment of chronic, moderate to severe cancer-related pain in terminally ill patients with a diagnosis of active cancer.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither the physician nor the patient knows the name of the assigned drug) study to evaluate the safety and effectiveness of JNJ-42160443 compared with placebo in the treatment of men and women 18 years of age or older who are terminally ill (ie, patients who are in or who are candidates for hospice or palliative [other medical care] care for end-of-life management) with moderate to severe, chronic, cancer-related pain that is not controlled by standard pain medications and who have a diagnosis of active cancer. The duration of the study will be approximately 62 weeks (includes screening, the 4-week double-blind phase followed by the 48-week open-label [study doctor and patient knows the name of the assigned treatment] extension phase and a posttreatment phase). A single dose of JNJ-42160443 or matching placebo given as an (subcutaneous [SC]) injection under the skin during the double-blind treatment period. During the open-label period, JNJ-42160443 will be given once every 4 weeks for up to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Terminally ill cancer patients as per judgment of the investigator (eg, patients who are in or who are candidates for hospice or palliative care for end-of-life management); Diagnosis of moderate to severe pain directly related to an active cancer that is not controlled by standard pain treatments.

Exclusion Criteria:Planned major surgical procedures during the double-blind treatment phase that may affect study outcomes; Prior treatment with any other investigational NGF inhibitor therapy; Known allergies, hypersensitivity, or intolerance to JNJ-42160443 or its excipients; Enrolled in any investigational study within the previous 4 weeks or 5 half-lives of the investigational drug (whichever is longer), or are currently enrolled in another investigational study at the time of screening

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The change in the average cancer-related pain intensity score. | From baseline (average cancer-related pain intensity score over the last 3 days before randomization) to the end of Week 4 (average cancer-related pain intensity score over the last 7 days of the double-blind treatment phase)

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | Up to Visit 10

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (40):
- United States (17):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Laguna Hills, California
  - Montebello, California
  - San Diego, California
  - Miami, Florida
  - Orlando, Florida
  - Stockbridge, Georgia
  - Anderson, Indiana
  - Lexington, Kentucky
  - Marrero, Louisiana
  - Shreveport, Louisiana
  - Farmington Hills, Michigan
  - Flat Rock, North Carolina
  - Cleveland, Ohio
  - Orem, Utah
  - Falls Church, Virginia
- France (5):
  - Lille
  - Lyon
  - Suresnes
  - Toulouse
  - Villejuif
- Poland (6):
  - Bygdoszcz
  - Gdansk
  - Gdansk-Zaspa
  - Lodz
  - Warsaw
  - Wroclaw
- Portugal (7):
  - Almada
  - Coimbra
  - Faro
  - Lisbon
  - Ponta Delgada
  - Porto
  - Setúbal
- Spain (5):
  - Barcelona
  - Madrid
  - Palma de Mallorca
  - San Sebastián de los Reyes
  - Terrasa Barcelona N/A